CLINICAL TRIAL: NCT00179244
Title: Risperidone vs. Bupropion ER Augmentation of SSRIs in Treatment-Resistant Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Principal Investigator, Richard C. Shelton, Director of Mood Disorder Clinic, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: RIS vs. BUP Augmentation Depr.; 040309
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Unipolar Depression
Keywords: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: Rispridone (drug) and Bupropion ER (drug)

SUMMARY:
The purpose of this study is to evaluate the comparative effectiveness of Risperdal (risperidone) or bupropion ER (extended release) combined with a SSRI medication and to test the relative safety of the combinations.

DETAILED DESCRIPTION:
Major depression is a severe disorder with serious consequences. Effective treatments are available; however, in clinical trials 30-40% of patients do not experience even a 50% reduction in depression severity scores, while 50-70% fail to achieve a full therapeutic response. Futhermore, impairment from the disorder continues essentially unabated in patients who are treated but do not fully remit. If anything, the situation is at least as bad or not worse in clinical practice. Clearly, alternatives are needed to manage this common clinical condition.

The addition of bupropion ER (extended release) to an SSRI has empirical support, and has become the most common augmentation strategy in the US. A comparative trial of the combination of risperidone or bupropion ER added to an SSRI in treatment resistant deperssion could help support risperidone for this condition; such a trial seems warranted at this time.

Patients who are currently on a SSRI at an adequate dosage for at least 3 weeks with no response, will be randomly assigned (open-label) to either risperidone or bupropion ER augmentation for a period of 6 weeks. Patients will be followed weekly at the beginning and bi-weekly towards the end of the trial to compare the response of each group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* DSM-IV diagnosis of major depressive disorder of at least moderate severity, but without psychotic features
* Ham-D 17 score of 18 or above
* Have a documentable history of 2 prior adequate trials of antidepressants including an SSRI without sufficient response. A clinically adequate trial is defined as having taken a minimum effective dose of an antidepressant for at least 3 weeks without a significant change in depressive symptoms.
* Must be currently on an serotonin uptake inhibitor (to include venlafaxine or duloxetine) at an adequate dose for at least 3 weeks.
* Ability and willingness to provide consent for participation in the study.

Exclusion Criteria:

* Any medical condition that would preclude treatment with an SSRI, risperidone, or bupropion ER
* Any clinically significant unstable medical condition
* Diagnosis of bipolar disorder or a primary diagnosis of any psychotic disorder
* Current psychotic symptoms (hallucination or delusions)
* Alcohol or drug abuse or dependence in the last 3 months (excluding nicotine and caffeine dependence/abuse) or abuse within the last month
* Documented non-response to the combination of a novel antipsychotic or bupropion ER and a SSRI
* Concomitant use of any psychotropic other than an SSRI or zolpidem (PRN for sleep)
* Score of 4 on the suicide item of the Ham-D scale and determination by the investigator of significant suicide risk
* Known sensitivity to risperidone or bupropion ER

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
MADRS (Montgomery Asberg's Depression Rating Scale)

SECONDARY OUTCOMES:
HAM-D(Hamilton Rating Scale for Depression ) 17-item
BDI (Beck Depression Inventory)
HAM-A (Hamilton Rating Scale for Anxiety)
Clinical Global Impression Scale and Severity and Improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Shelton, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States